CLINICAL TRIAL: NCT04768686
Title: A Phase 2 Study to Assess the Safety, Efficacy of FLX475 Combined With Pembrolizumab in Patients With Advanced or Metastatic Gastric Cancer
Brief Title: FLX475 Combined With Pembrolizumab in Patients With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-CCRI-201; KEYNOTE-B83 (Other: Merck Sharp & Dohme LLC); MK-3475-B83 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FLX475 and pembrolizumab combination therapy (Experimental): * Cohort 1: EBV negative / CPI naïve gastric cancer patient who has had a disease progression after at least 2 prior systemic treatments for advanced or metastatic gastric cancer
  * Cohort 2: EBV positive / CPI naïve gastric cancer patient (as determined by standard methods, e.g. EBER ISH or LMP-1 IHC) who had at least 1 prior systemic treatment for advanced or metastatic gastric cancer
  Interventions: Drug: FLX475; Drug: Pembrolizumab

INTERVENTIONS:
Drug: FLX475 — tablet
Drug: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®

SUMMARY:
This clinical study is a Phase 2, open-label study to assess the efficacy, safety profile of FLX475 combined with pembrolizumab in patients with advanced or metastatic gastric cancer. This study is designed to assess the potential anti-tumor activity when administered at the 100mg QD of FLX475 with pembrolizumab and will be conducted (2) cohorts as detailed below.

* Cohort 1: EBV negative / CPI naïve gastric cancer subjects who have progressed on at least 2 prior systemic treatments for advanced or metastatic gastric cancer
* Cohort 2: EBV positive / CPI naïve gastric cancer subjects who had at least 1 prior systemic treatment for advanced or metastatic gastric cancer

Approximately 90 subjects may be enrolled across two cohorts to examine the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed, advanced, relapsed or metastatic gastric or gastroesophageal junction adenocarcinoma
* Patient must have one of the following diagnoses to be eligible for enrollment into cohorts:

  * Cohort 1: Checkpoint inhibitor naïve Epstein-Barr Virus negative (EBV-) gastric cancer patient who has had a disease progression after at least 2 prior systemic treatments for advanced or metastatic gastric cancer
  * Cohort 2: Checkpoint inhibitor naïve Epstein-Barr virus positive (EBV+) gastric cancer patient (as determined by standard methods, e.g. EBER ISH or LMP-1 IHC) who had at least 1 prior systemic treatment for advanced or metastatic gastric cancer
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Patient must have at least one measurable lesion at baseline by computed tomography(CT) or magnetic resonance imaging (MRI)
* Tumor available for biopsy

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137), any history of discontinuing from that treatment due to Grade 3 or higher immune-related adverse event (irAE)
* Patient with MSI-H status
* Active autoimmune disease or serious autoimmune disease within past 2 years requiring systemic therapy
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, (non-infectious) pneumonitis that required steroids, or clinical symptoms of active pneumonitis
* Significant cardiovascular disease. New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, or chronic Grade 3 hypertension.
* Significant screening electrocardiogram (ECG) abnormalities
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Hanllym University Medical Center, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening will occur from Day -30 to Day -1. Once screening procedures are completed and eligibility is confirmed, subjects will be enrolled for the study and start study treatment. There is no pre-assignment planned.
Groups:
- FLX475 and Pembrolizumab Combination Therapy: * Cohort 1: EBV negative / CPI naïve gastric cancer patient who has had a disease progression after at least 2 prior systemic treatments for advanced or metastatic gastric cancer
  * Cohort 2: EBV positive / CPI naïve gastric cancer patient (as determined by standard methods, e.g. EBER ISH or LMP-1 IHC) who had at least 1 prior systemic treatment for advanced or metastatic gastric cancer
  FLX475: tablet
  Pembrolizumab: IV infusion
Period: Overall Study
Arm/Group | FLX475 and Pembrolizumab Combination Therapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of FLX475 or pembrolizumab. All demographics, Baseline characteristics, efficacy and safety data were analyzed using the Treated Set as a primary analysis population.
Arm/Group | FLX475 and Pembrolizumab Combination Therapy
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years] — Population: This clinical trial was designed with two separate cohorts. The overall baseline population was based on the total treated set across both cohorts, while the results for age were reported separately for each cohort (10 patients each).
  years
    Total | 64.5 [44 to 80]
    Cohort 1: number analyzed (Participants) | 10
    Cohort 1 | 60.0 [44 to 80]
    Cohort 2: number analyzed (Participants) | 10
    Cohort 2 | 65.5 [52 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This clinical trial was designed with two separate cohorts. The overall baseline population was based on the total treated set across both cohorts, while the results for sex were reported separately for each cohort (10 patients each).
  Participants
    Total: Female | 5
    Total: Male | 15
    Cohort 1: number analyzed (Participants) | 10
    Cohort 1: Female | 3
    Cohort 1: Male | 7
    Cohort 2: number analyzed (Participants) | 10
    Cohort 2: Female | 2
    Cohort 2: Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This clinical trial was designed with two separate cohorts. The overall baseline population was based on the total treated set across both cohorts, while the results for race/ethnicity were reported separately for each cohort (10 patients each).
  Participants
    Total: Asian | 20
    Total: Other | 0
    Cohort 1: number analyzed (Participants) | 10
    Cohort 1: Asian | 10
    Cohort 1: Other | 0
    Cohort 2: number analyzed (Participants) | 10
    Cohort 2: Asian | 10
    Cohort 2: Other | 0
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] — Population: This clinical trial was designed with two separate cohorts. The overall baseline population was based on the total treated set across both cohorts, while the results for baseline height were reported separately for each cohort (10 patients each).
  cm
    Total | 165.31 (8.16)
    Cohort 1: number analyzed (Participants) | 10
    Cohort 1 | 163.93 (8.94)
    Cohort 2: number analyzed (Participants) | 10
    Cohort 2 | 166.68 (7.51)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] — Population: This clinical trial was designed with two separate cohorts. The overall baseline population was based on the total treated set across both cohorts, while the results for BMI were reported separately for each cohort (10 patients each).
  kg/m2
    Total | 21.67 (3.77)
    Cohort 1: number analyzed (Participants) | 10
    Cohort 1 | 21.94 (2.75)
    Cohort 2: number analyzed (Participants) | 10
    Cohort 2 | 21.39 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The primary efficacy endpoint is Objective Response Rate (ORR) defined as the proportion of subjects whose confirmed best overall response is either Complete Response (CR) or Partial Response (PR) according to RECIST version 1.1. For the efficacy endpoints (such as ORR and DCR), frequency and percentage of subjects who have achieved a response will be summarized by cohort and 95% 2-sided confidence interval will be calculated by Clopper-Pearson method.
Time Frame: Initial assessment performed after the first 2 cycles, then every 2 cycles for the first year, followed by every 3 cycles thereafter for up to 2 years and at any time per investigator's discretion and at ED/EOT, up to 2 years.
Population: The treated set included all subjects who received at least 1 dose of FLX475 or pembrolizumab. All demographics, Baseline characteristics, efficacy and safety data were analyzed using the Treated Set as a primary analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: EBV Negative / CPI naïve Gastric Cancer: ◦ Cohort 1: EBV negative / CPI naïve gastric cancer patient who has had a disease progression after at least 2 prior systemic treatments for advanced or metastatic gastric cancer
- Cohort 2: EBV Positive / CPI naïve Gastric Cancer: ◦ Cohort 2: EBV positive / CPI naïve gastric cancer patient (as determined by standard methods, e.g. EBER ISH or LMP-1 IHC) who had at least 1 prior systemic treatment for advanced or metastatic gastric cancer
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 10 | 10
percentage of participants | 0 [0 to 30.8] | 60.0 [26.2 to 87.8]

2. Secondary Outcome: Disease Control Rate (DCR) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The Disease Control Rate (DCR) is defined as the proportion of subjects with confirmed best overall response of CR, PR or SD according to RECIST version 1.1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 10 | 10
percentage of participants | 20.0 [2.5 to 55.6] | 60.0 [26.2 to 87.8]

3. Secondary Outcome: Time to Response (TTR) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The Time to Response (TTR) is defined as the time from the date of first administration of study treatment to first documented Complete Response (CR) or Partial Response (PR).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 10 | 10
months | NA [NA to NA] — Not available due to no responder. | 2.7 [1.2 to NA] — Not estimable due to insufficient events near the median.

4. Secondary Outcome: Duration of Response (DoR) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The Duration of Response (DoR) is measured from the date of the first observation of tumor response (Complete Response (CR) or Partial Response (PR), whichever occurs first) to the date of disease progression or death for the subject with an objected response.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 0 | 6
months |  | 17.3 [2.7 to NA] — Not estimable due to insufficient events near the median.

5. Secondary Outcome: Progression-free Survival (PFS) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The Progression-free Survival (PFS) is defined as the time from the date of first administration of study treatment to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 10 | 10
months | 1.4 [1.1 to 1.5] | 10.4 [1.0 to NA] — Not estimable due to insufficient events near the median.

6. Secondary Outcome: Overall Survival (OS) in Subjects Treated With FLX475 in Combination With Pembrolizumab
Description: The Overall Survival (OS) is defined as the duration of time from the treatment start date to time to death from any cause. If subjects survive at the time of analysis, the subject will be censored at the last date of survival confirmed.
Time Frame: From baseline (Cycle 1 Day 1 prior to administration of the first study dose) until death from any cause.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
Number analyzed (Participants) | 10 | 10
months | 7.5 [1.4 to NA] — Not estimable due to insufficient events near the median. | NA [2.3 to NA] — Not estimable due to insufficient events.

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events were recorded and followed through 30 days following cessation of study treatment (or 30 days after final dose if new anticancer therapy initiates), or until resolution, whichever comes first, up to 27 months. All Serious Adverse Events (SAEs) were reported after the consent form is signed through 90 days following cessation of study treatment, or 30 days after final dose if the subject initiates new anticancer therapy, whichever occurs first, up to 27 months.
Description: Safety endpoints were analyzed using the Treated Set. All AEs were coded using MedDRA Version 26.1 and graded using NCI-CTCAE Version 5.0. All AE summaries were restricted to treatment-emergent adverse events (TEAEs) only.
Arm/Group | Cohort 1: EBV Negative / CPI naïve Gastric Cancer | Cohort 2: EBV Positive / CPI naïve Gastric Cancer
All-Cause Mortality (participants affected / at risk) | 3/10 | 4/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 5/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: EBV Negative / CPI naïve Gastric Cancer (N=10) | Cohort 2: EBV Positive / CPI naïve Gastric Cancer (N=10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Internal hernia (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: EBV Negative / CPI naïve Gastric Cancer (N=10) | Cohort 2: EBV Positive / CPI naïve Gastric Cancer (N=10)
Electrocardiogram QT prolonged (Investigations) | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Asthenia (General disorders) | 0 | 3
Fatigue (General disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2
Lipase increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Amylase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Internal hernia (Gastrointestinal disorders) | 0 | 1
Malignant ascites (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive coug (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Retinopathy (Eye disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT04768686/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04768686/SAP_001.pdf